CLINICAL TRIAL: NCT04445220
Title: A Multi-center, Randomized, Case Controlled, Double-blind, Ascending-dose Study of Extracorporeal Mesenchymal Stromal Cell Therapy (SBI-101 Therapy) in COVID-19 Subjects With Acute Kidney Injury Receiving Renal Replacement Therapy
Brief Title: A Study of Cell Therapy in COVID-19 Subjects With Acute Kidney Injury Who Are Receiving Renal Replacement Therapy
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Sentien Biotechnologies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SBI-101-02
Record Dates: First submitted 2020-06-22; First posted 2020-06-24 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2021-08

CONDITIONS: COVID-19; Acute Kidney Injury; Sepsis
Keywords: CRRT; AKI; Continuous renal replacement therapy; MSC; Mesenchymal stromal cells; Mesenchymal stem cells; Stem cells; Cell therapy
MeSH Terms: conditions — COVID-19; Acute Kidney Injury; Sepsis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose cohort (Experimental): SBI-101 device containing 250 million MSCs
  Interventions: Biological: SBI-101
- High dose cohort (Experimental): SBI-101 device containing 750 million MSCs
  Interventions: Biological: SBI-101
- Case controls (No Intervention): Case control subjects will receive only standard-of-care treatment and will be followed for the same safety assessments as active study participants.

INTERVENTIONS:
Biological: SBI-101 — SBI-101 is a biologic/device combination product that combines two components: allogeneic human mesenchymal stromal cells (MSCs) and an FDA-approved plasmapheresis device. SBI-101 is administered via integration into a Continuous Renal Replacement Therapy circuit and is designed to regulate inflammation and promote repair of injured tissue.
  Arms: High dose cohort; Low dose cohort

SUMMARY:
The purpose of this study is to assess the safety and tolerability of the investigational product, SBI-101, in subjects with an infectious etiology of Acute Kidney Injury (AKI). SBI-101 is a biologic/device combination product designed to regulate inflammation and promote repair of injured tissue using allogeneic human mesenchymal stromal cells. SBI-101 will be integrated into the renal replacement circuit and patients will be treated for up to 24 hours.

ELIGIBILITY:
Inclusion Criteria:

* Documented evidence of infection, e.g., positive PCR for COVID-19, positive blood cultures for systemic infection, active urinary sediment to suggest UTI, or any imaging supportive of a clinical diagnosis of infection, for example, pulmonary infiltrate on chest x-ray to suggest pneumonia, pancreatitis on CT imaging, abdominal collection, etc.
* AKI as determined by the Investigator based on his/her clinical judgment
* Receiving or planned to receive RRT in < 24 hours
* Able to tolerate indwelling intravascular access
* Has tolerated CRRT for at least 6 hours prior to IP treatment
* Have maintained hemodynamic stability for at least 6 hours prior to IP treatment with only minor changes in pressure support medication required (if used)
* Vascular access (catheter placement) is patent and capable of supporting CRRT for the duration of IP treatment
* Likely to require RRT for at least an additional 48 hours
* Potassium level >3.6 and <5.5 mEq/L or >3.6 and < 5.5 mmol/L prior to IP treatment
* SaO2 > 92% prior to IP initiation
* Blood pH > 7.2 prior to IP initiation
* Medically cleared to receive anticoagulation per institutional standard of care / PI prescribed protocol and meeting protocol defined anticoagulation targets prior to receipt of IP
* Ability to give informed consent or have a legally authorized representative do so

Exclusion Criteria:

* Female subjects who are pregnant, planning to become pregnant, or lactating
* MAP <70 mmHg immediately prior to IP initiation
* Systolic blood pressure < 90 mmHg immediately prior to IP initiation
* Mechanical ventilator support requiring FiO2 > 80% prior to IP initiation
* Receiving extracorporeal membrane oxygenation (ECMO)
* Liver disease with Child Pugh score of > 7 prior to IP initiation
* High sensitivity cardiac Troponin level (hs-cTn) > 100.0 ng/L prior to IP initiation or other equivalent Troponin test result prior to IP initiation
* Hepatorenal syndrome
* AKI due to post-renal outflow obstruction
* Acute or chronic vasculitis of any etiology
* Chronic systemic infection
* Subjects with a past medical history of an inherited or acquired hypercoagulable condition independent of COVID-19
* Patients with a past medical history of an allergic response to MSC therapy
* Participation in another interventional trial with the exception of studies of antivirals, corticosteroids, hydroxychloroquine, azithromycin, or angiotensin converting enzyme inhibitors/angiotensin receptor blockers (or related compounds)
* Active malignancy(-ies) and/or receiving active treatment for a malignancy(-ies), with the exception of non-melanoma skin cancer
* Subjects, who in the opinion of the Investigator, are likely to require escalating doses of vasopressors to attain and/or maintain hemodynamic stability, or subjects who have reached the institutionally defined maximum level of vasopressor support within 12 hours of intended IP integration
* Imminent death in <24 hours
* Organ failure affecting more than 2 non-renal organs
* Platelet count <50,000/μL or other serious hematological abnormalities that would place subject in imminent danger of death
* Lactate levels >8 mmol/L suggestive of severe end-organ hypoperfusion prior to the time of IP integration
* Any prior medical condition or recent surgical procedure, planned significant medical interventions or procedures that, in the judgment of the Investigator, would prevent the subject from safely participating in and/or completing all study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2020-11-19 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-09 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability as measured by incidence of IP-related serious adverse events | Outcomes and Serious Adverse Events through Day 180

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - Medical University of South Carolina, Charleston, South Carolina

IPD SHARING:
Plan to Share IPD: No